CLINICAL TRIAL: NCT04938999
Title: Effects of a Music-visual Guided Physical Activity Promotion Program Among Adults With Intellectual Disability Living in Residential Care Facilities: A Cluster-randomized Controlled Trial
Brief Title: Music-visual Guided Physical Activity Promotion for Adults With Intellectual Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Ho Yu CHENG, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019.624
Record Dates: First submitted 2021-06-13; First posted 2021-06-25 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Intellectual Disability
Keywords: physical activity; residential care; information-motivation-strategy model
MeSH Terms: conditions — Intellectual Disability; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Eligible participants recruited from the same facility will be allocated to either intervention or control groups accordingly. Group allocation will be concealed from outcome assessors and made according to the random group allocation sequence generated by an independent statistician and the sequence of entry into the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MVgPA group (Experimental): The MVgPA group consists of 24 sessions conducted over 12 weeks for the study participants by the staff of residential care facilities.
  The structured MVgPA group session (10 - 12 participants) will be conducted twice per week. The 75-min music-paced physical activities will be presented in the PowerPoint slideshow. The instructions for an upper limb exercise will be presented in a large number pad in the slideshow, and the participants will then be asked to follow the actions and directions presented on the slide.
  Interventions: Behavioral: Music-visual guided physical activity (MVgPA)
- Control group (Other): residential care facilities will conduct their usual activities during the study period. A trained RA2 will record the activities conducted by the residential care facilities during the study period.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Music-visual guided physical activity (MVgPA) — The MVgPA adopts the information-motivation-strategy model to address the personal and environmental challenges in PA initiation and maintenance of adults with intellectual disability.
  To support the staff of residential care facilities in implementing 24 sessions of MVgPA in 12 weeks, the first six sessions will be led by the RA1 and co-facilitated by the staff, while the subsequent sessions will be conducted by the staff only. At week 6, another set of MVgPA will be implemented to increase the participant's interest; two sessions will be co-facilitated by RA1. At weeks 6 and 9, the RN and RA1 will hold a meeting with the staff of the residential care facilities to acknowledge the achievement of the staff and adults with ID, as well as to address any of their concerns related to the implementation of MVgPA, and to identify the facilitators and tackle barriers to the implementation of the MVgPA.
  Arms: MVgPA group
Behavioral: Usual care — As control group, residential care facilities will conduct their usual activities during the study period. A trained RA will record the activities conducted by the residential care facilities during the study period.
  Arms: Control group

SUMMARY:
Objective: Although physical activity (PA) is cardiometabolic and psychologically beneficial to adults with intellectual disability (ID), its initiation and maintenance remain problematic. We examine the effects of a music-visual guided PA (MVgPA) intervention on the PA level, PA self-efficacy and interest as well as functional exercise capacity of adults with ID.

Hypothesis: Compared with usual care, MVgPA can significantly increase the participant's PA level and improve their PA self-efficacy and interest, and functional exercise capacity.

Design and participants: This cluster-randomized controlled trial will recruit 400 Chinese adults with mild to moderate ID from 20 residential care facilities.

Intervention: Based on the information-motivation-strategy model, MVgPA comprises a motivational and strategical preparatory session and ongoing support to residential service providers and a 12-week group-based staff-facilitated MVgPA (two 75-min session/week) for adults with ID. Outcome measurement PA level (primary outcome) will be measured by using an activity tracker. PA self-efficacy and interest will be measured by the Baseline Interview Questionnaire and visual analogue scale respectively. Functional exercise capacity will be measured by six-minute walk test. All outcomes will be measured at baseline, 13 and 25 weeks.

Data analysis: Intervention effects will be estimated using three-level mixed effects model.

Expected results: MVgPA will effectively enhance the PA levels of adults with ID. After intervention implementation, we expect that at least 50% of the residential care facilities allocated to the intervention group will demonstrate their willingness to continue to implement the MVgPA program (score 4 out of 6, 6 = most willing).

DETAILED DESCRIPTION:
The specific objectives of this project are to (1) evaluate the effectiveness of this intervention in improving the PA level of these adults, enhancing their self-efficacy and interest in performing PA and improving their functional exercise capacity by conducting a cluster-randomized controlled trial, and (2) examine the acceptability of this intervention among the participants and the staff of residential care facilities.

Participant recruitment The person-in-charge of residential care facilities and the non-governmental organizations that serve adults with ID, including the Hong Chi Association who had collaborated with us in our pilot project, will be approached by the research team to seek their collaboration and support in recruiting participants and implementing the project. The research team will organize promotion talks and distribute promotion leaflets of the project to potential participants and their families or legal guardians. To ensure safety of the participants, PA pre-participation health screening will be performed in accordance with the guidelines of American College Sport Medicine. Medical clearance/approval to participate MVgPA will be sought if they have known cardiovascular, metabolic and/or renal disease, or signs and symptoms suggesting these diseases (as detailed in Appendix 1). An information sheet related to the MVgPA, including the heart rates during the PA and type of exercise, will be provided to the physicians.

Sample size calculation A similar study for adults with ID in community residences showed an effect size of 0.35 on PA level change. Assuming a similar effect size on PA level change in our proposed trial, a sample size of 129 participants per each of the control and intervention groups will provide the study with 80% power at 2-sided 5% level of significance, as estimated using the power analysis software PASS 13.0 (NCSS, Kaysville, USA). Furthermore, to account for potential reduction in statistical efficiency due to randomization by residential care facilities (clusters) instead of individual participants, a variance inflation factor, called design effect, will be applied to impose to the estimated sample size. The design effect is given by 1 + (m-1)*ICC, where m=average cluster size and ICC=intracluster correlation coefficient of the underlying outcome. We anticipate that the outcomes of the participants recruited from the same residential care facility are unlikely correlated with one another, particularly for the PA outcome. In this regard, the ICC would be small. A synthesis study revealed that ICC tends to be small in primary care research with a median of 0.005 and inter-quartile range of 0.000 to 0.021. Allowing for a conservative ICC of 0.01 in our proposed study, at least 16 participants per each of the 20 residential care facility are therefore required. Furthermore, to allow up to 20% attrition rate, at least 20 participants per facility will be recruited.

Cluster randomization Randomization will be performed at the cluster level (residential care facility) instead of individual participants to avoid contamination between the intervention and control groups. The facilities will be randomized to either intervention or control group in a 1:1 ratio. Eligible participants recruited from the same facility will be allocated to either intervention or control groups accordingly. Group allocation will be concealed from outcome assessors and made according to the random group allocation sequence generated by an independent statistician and the sequence of entry into the study.

Data analysis By considering the potential design effect of the randomization conducted in cluster level instead of individual participants, the outcome analysis will be performed on the basis of a three-level mixed effects model accounting for inter-correlation among individuals within the same cluster as well as intra-correlation over time within an individual and variations between individuals. This type of model can account for intra-correlated clustered and repeated measures data and produce unbiased estimates even in the presence of missing data, provided that the data are missing at random. Mixed-effects model will be used to compare the differential changes in each outcome variables (PA level, PA self-efficacy and interest, and exercise capacity) across time (T0, T1, T2) between the two groups. Positive significant group-by-T1 and group-by-T2 interaction-terms in the mixed-effects models indicate significantly greater increment of intervention group in the underlying outcome than the control group at the respective time-points with respect to T0.

ELIGIBILITY:
Inclusion Criteria:

* Chinese adults who are aged 18 years to 64 years and are diagnosed with mild or moderate ID based on the information provided by the residential care facilities;
* Able to understand basic information and instructions of the intervention and to make decisions upon their participation;
* Classified as physically inactive (i.e., <150-min moderate-intensity or 75-min vigorous-intensity PA/week);
* Currently using residential service user as stated in the Social Welfare Department of Hong Kong SAR.

Exclusion Criteria:

* Currently enrolled in a regular exercise program;
* Physically unable to participate in the MVgPA, such as having significant mobility problem;
* Participation to MVgPA will put them at physiological risk; or
* At risk of self-harm as determined by the staff of the residential care facilities.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
PA level | Change from baseline PA level at one-week and three-month post-intervention
  The physical activity level of participants will be assessed in terms of minutes of moderate-to-vigorous PA by using an activity tracker

SECONDARY OUTCOMES:
Self-efficacy of performing physical activity (PA self-efficacy) | Change from baseline PA self-efficacy level at one-week and three-month post-intervention
  Self-efficacy of performing physical activity will be measured by using the Chinese version of the self-efficacy scale of the baseline interview questionnaire
Functional exercise capacity | Change from baseline functional exercise capacity at one-week and three-month post-intervention
  6 minutes walk test

OTHER OUTCOMES:
Interest in performing physical activity and satisfaction level of the participants of intervention group | one-week post-intervention
  a visual analogue scale, which consists of a 100 mm long line with the left anchor representing "0 = no interest/not satisfied at all" and the right anchor representing "100 = most interested/most satisfied"
satisfaction of residential service providers with the intervention and their willingness to continue with the program | one-week post-intervention
  author-developed questionnaire (score 0 = not satisfied at all/unwilling to continue with the program; 5 = most satisfied/will continue with the program for sure)

CONTACTS AND LOCATIONS:
Locations (1):
- The Nethersole School of Nursing, Chinese University of Hong Kong, Hong Kong, Please Select, China

IPD SHARING:
Plan to Share IPD: No